CLINICAL TRIAL: NCT03388177
Title: Yoga-based Therapy for Young Women With Depression: a Randomized Controlled Trial
Brief Title: Yoga for Young Women With Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Groningen (Other)
Collaborators: Lentis Psychiatric Institute (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Triodos Foundation (Unknown)
Responsible Party: Principal Investigator, Brian Ostafin, Associate Professor, University of Groningen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 60-63600-98-127
Record Dates: First submitted 2017-11-02; First posted 2018-01-02 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Young adult women; Yoga
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The project uses a blinded rater to assess the primary outcome measure of symptoms of depression
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual + Yoga-based therapy (Experimental): The yoga-based therapy (YBT) group will receive YBT in addition to treatment-as-usual (TAU). YBT will be administered with a manualized protocol and delivered in a group format consisting of nine weekly sessions of 1,5 hours. Group sessions consist of hatha yoga practices of physical postures, breathing practices, and meditation. Each session has a different theme. The practices will primarily consist of yoga exercises (80%) and meditation (e.g., breathing practices) (20%). Between sessions, participants complete an online module with additional psychoeducation and a practice video to encourage home practice for 30-45 minutes a day. YBT will be delivered by a psychologist who is also a trained yoga teacher.
  Interventions: Behavioral: Yoga-based therapy; Other: Treatment as usual
- Treatment as usual (Other): The treatment as usual (TAU)-only condition will consist of interventions recommended by the Dutch guidelines for depression. These include the combination of pharmacotherapy (antidepressant medications) and psychotherapy (e.g., cognitive behavioral therapy [CBT], interpersonal psychotherapy). Lentis mental health clinicians will administer TAU. In order to improve ability to interpret study results, the investigators will record frequency, content (e.g., cognitive restructuring), format (group versus individual), and intensity of contact within TAU. Such quantification of TAU will allow us to address alternative explanations (e.g., contact time) in the case of positive results for YBT.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Yoga-based therapy
  Arms: Treatment as usual + Yoga-based therapy
Other: Treatment as usual
  Other Names: Care as usual

SUMMARY:
The investigators examine whether adding yoga-based therapy (YBT) to treatment as usual (TAU) for young adult women (age 18-34 years) with a primary diagnosis of MDD leads to (1) greater reductions in symptoms and (2) greater cost-effectiveness in that the economic benefits of adding YBT to TAU outweigh the costs.

DETAILED DESCRIPTION:
BACKGROUND Major Depressive Disorder (MDD) is widespread, as nearly one in five Dutch will experience the disorder within their lifetime. In addition to individual suffering, MDD creates great economic costs in the Netherlands and is a leading contributor to the national disease burden. Although first-step interventions can be helpful, many individuals with MDD do not seek treatment and current interventions often fail to prevent the development of chronic, relapsing MDD. There is thus a pressing need to develop and test new interventions for depression. This need is particularly urgent in young adult women, as this population is especially vulnerable to developing MDD. Yoga-based interventions represent an innovative approach with great potential for treating depression. The rationale of using yoga as a MDD intervention in young women includes initial findings that yoga reduces depressive affect and yoga's appeal in this population. Although the initial findings are promising, previous research has a number of methodological limitations such as insufficient statistical power, and short follow-up periods. The proposed project is designed to use rigorous methods to examine yoga as a treatment for acute depression and as means of preventing the transition to a chronic, relapsing disorder in a sample of young women.

OBJECTIVE The overall objective of this project is to examine the potential benefits of adding a yoga-based intervention (YBI) to treatment as usual (TAU) for young women with major depressive disorder (MDD). This objective will be examined with the following four specific aims: (1) to examine whether adding YBI to TAU leads to greater and sustained reductions in symptoms, and (2) better general functioning in young women with MDD at post-intervention and at 6- and 12-month follow-up, (3) to examine the cost-effectiveness of adding YBI to TAU and, (4) these effects are mediated by change in rumination, self-criticism, intolerance of uncertainty, interoceptive awareness, and dispositional mindfulness.

HYPOTHESES The hypotheses (H) are that compared to TAU, YBI+TAU will lead to: (H1) greater reductions in depressive symptoms, assessed with clinician-administered and self-report measures, and (H2) better general functioning, defined as (H2.1) daily functioning, (H2.2) quality of life and physical health, and (H2.3) positive psychological functioning. The investigators further hypothesize that (H4) compared both to TAU, YBT (+TAU) will show greater cost-effectiveness, and that these YBI effects on symptoms of depression are partially mediated by (H4.1) reduced self-report and implicit rumination about the causes and consequences of negative events and moods, (H4.2) reduced self-report and implicit self-criticism/increased self-compassion after perceived failures, (H4.3) decreased intolerance of uncertainty, (H4.4) increased body awareness/interoceptive awareness, and (H4.5) increased mindfulness.

STUDY DESIGN The study will consist of a randomized controlled trial comparing YBT+TAU with TAU. Assessments are completed at pre- and post-intervention (or equivalent time period in TAU), and at 6- and 12-month follow-up.

STUDY POPULATION Young adult women (age 18-34 years) with a primary diagnosis of MDD.

INTERVENTION The intervention will consist of manualized YBT administered in 9 weekly 90-minute group sessions with home practice +TAU.

USUAL CARE TAU will consist of interventions recommended by the Dutch guidelines for depression, including psychotherapy, pharmacotherapy, psychosocial support by psychiatric nurses, or some combination of these.

OUTCOME MEASURES Primary outcome measures will consist of clinician-administered and self-report measures of depression symptoms and the presence/absence of a diagnoses of Major Depressive Disorder. Secondary outcome measures are daily functioning, quality of life and physical health, and positive psychological functioning. Potential mediators are self-report measures of perseverative thinking, self-criticism, intolerance of uncertainty, interoceptive awareness and dispositional mindfulness, and implicit measures of perseverative thinking and self-criticism. Quality-Adjusted Life Years will be used as primary outcome measure in the economic analysis.

SAMPLE SIZE/DATA ANALYSIS A sample of N=64/group will be recruited in order to have power of 80% (alpha=.05) to detect medium effect size differences between groups. Allowing attrition of 25%, 170 (85/group) patients will be recruited. Repeated-measures ANOVAs and Chi-square analyses will be conducted.

COST EFFECTIVENESS ANALYSIS An economic evaluation will be conducted alongside the clinical study to assess the potential cost-effectiveness of YBT compared to TAU from a societal perspective. A budget impact analysis (BIA) will be conducted to inform decision-makers about the potential financial consequences of the adoption and diffusion of YBT in the Dutch healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of a major depressive disorder.
* Age ≥ 18 and ≤ 34.
* Ability to fluently read, write, and speak Dutch.

Exclusion Criteria:

* Current diagnoses of bipolar disorder and substance dependence.
* Current psychotic symptoms.
* Active suicidality.
* Unwilling or inability to attend to 9 weekly sessions of yoga.
* Regular yoga practice (on average over the past 6 months, 30 or more minutes per week).

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Estimated)
Dates: Start 2016-12-16 (Actual); Primary Completion 2018-12-16 (Estimated); Study Completion 2019-12-16 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scales (from baseline to 10-15 weeks post baseline, 6-month follow-up and 12-month follow-up) | Baseline, 10-15 weeks post baseline, 6 and 12 months follow-up
  Clinician-administered. Hamilton Depression Rating Scales: to assess symptoms of depression; total scores from 0-52; higher value represent more symptoms of depression.
Change in Depression scale of Depression Anxiety Stress Scales (from baseline to 10-15 weeks post baseline, 6-month follow-up and 12-month follow-up) | Baseline, 10-15 weeks post baseline, 6 and 12 months follow-up
  Self-report. Depression Anxiety Stress Scales: to assess symptoms of depression with total possible score of 0-21; higher values represent more depression

SECONDARY OUTCOMES:
Structured clinical interview for DSM-IV | 12 months follow-up
  Clinician administered. Structured clinical interview for DSM-IV to assess diagnosis of MDD; 5 out of 9 symptoms to have a diagnosis of MDD.
Change in Anxiety scale of Depression Anxiety Stress Scales (from baseline to 10-15 weeks post baseline, 6-month follow-up and 12-month follow-up) | Baseline, 10-15 weeks post baseline, 6 and 12 months follow-up
  Self-report. Depression Anxiety Stress Scales: to assess symptoms of anxiety with total possible score of 0-21; higher values represent more anxiety
Change in Stress scale of Depression Anxiety Stress Scales (from baseline to 10-15 weeks post baseline, 6-month follow-up and 12-month follow-up) | Baseline, 10-15 weeks post baseline, 6 and 12 months follow-up
  Self-report. Depression Anxiety Stress Scales: to assess symptoms of stress with total possible score of 0-21; higher values represent more stress
Healthcare use with healthcare consumption scale (from baseline to 10-15 weeks post baseline, 6-month follow-up and 12-month follow-up) | Baseline, 10-15 weeks post baseline, 6 and 12 months follow-up
  The healthcare consumption scale is modified from the Trimbos/iMTA questionnaire for costs associated with psychiatric illness (TiC-P). Societal costs will be calculated by combining results of the healthcare consumption scale with cost prices per unit of healthcare used.
Health-related quality of life with EQ-5D-5L (from baseline to 10-15 weeks post baseline, 6-month follow-up and 12-month follow-up) | Baseline, 10-15 weeks post baseline, 6 and 12 months follow-up
  The EQ-5d-5L is a preference-based health instrument aimed at 5 health dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each can be scored at 5 levels (ranging from no problems to extreme problems). In the context of cost-effectiveness studies, results of the EQ-5D-5L can be used to assess QALYs (when combined with information on life years).
Change in Perseverative thinking Questionnaire (from baseline to 10-15 weeks post baseline, 6-month follow-up and 12-month follow-up) | Baseline, 10-15 weeks post baseline, 6 and 12 months follow-up
  Self report. To assess repetitive negative thinking; total scores from 0-60; higher values represent more repetitive negative thinking.
Change in Exogenous cuing task (from baseline to 10-15 weeks post baseline) | Baseline and 10-15 weeks post baseline
  This is a reaction time task that assesses attentional bias to depression-related stimuli. Larger difference score values (responses to depression-related vs. neutral stimuli) indicate greater automatic orienting to and greater difficulty in disengaging from depression-related stimuli.
Change in Self-Compassion Scales (from baseline to 10-15 weeks post baseline, 6-month follow-up and 12-month follow-up) | Baseline, 10-15 weeks post baseline, 6 and 12 months follow-up
  Self report. Self-Compassion Scales used to assess self-compassion; total scores from 24-168, 6 subscales from 4-28; higher values represent more self-compassion; subscales are averaged as well as the total score (so scores range from 1-7).
Change in Implicit Association Test (of depression self-concept) (from baseline to 10-15 weeks post baseline) | Baseline and 10-15 weeks post baseline
  The Implicit Association Test is a reaction time task that will be used to assess the strength of associations between the categories of 'self' and 'depression' (relative to 'other' and 'elated'.
Change in Intolerance of Uncertainty Scale-short form (from baseline to 10-15 weeks post baseline, 6-month follow-up and 12-month follow-up) | Baseline, 10-15 weeks post baseline, 6 and 12 months follow-up
  Intolerance of Uncertainty Scale-short form: to assess intolerance of uncertainty; total scores from 12-60; higher values represent more intolerance of uncertainty.
Change in Five-Facet Mindfulness Questionnaire-short form (from baseline to 10-15 weeks post baseline, 6-month follow-up and 12-month follow-up) | Baseline, 10-15 weeks post baseline, 6 and 12 months follow-up
  Self report. Five-Facet Mindfulness Questionnaire-short form: to assess dispositional mindfulness; total scores from 24-120, 5 subscales from 4/5-20/24 (1 subscale consists of 4 items, the others of 5); higher scores represent more mindfulness; subscales are summed to combine for total score
Change in Awareness scale of the Scale of Body Connection (from baseline to 10-15 weeks post baseline, 6-month follow-up and 12-month follow-up) | Baseline, 10-15 weeks post baseline, 6 and 12 months follow-up
  Self-report (Awareness scale of the Scale of Body Connection)
Change in Work and Social Adjustment Scale (from baseline to 10-15 weeks post baseline, 6-month follow-up and 12-month follow-up) | Baseline, 10-15 weeks post baseline, 6 and 12 months follow-up
  Self-report. Work and Social Adjustment Scale: to assess work and social functioning; total scores from 0-40; higher values represent more problems in work and social functioning.
Change in World Health Organization Quality of Life Questionnaire-brief (from baseline to 10-15 weeks post baseline, 6-month follow-up and 12-month follow-up) | Baseline, 10-15 weeks post baseline, 6 and 12 months follow-up
  World Health Organization Quality of Life Questionnaire-brief: to assess quality of life; total scores from 25-125, 5 subscales from 2-10 (1 subscale contains 2 items), 7-35 (1 subscale contains 7 items), 6-30 (1 subscale contains 6 items), 3-15 (1 subscale contains 3 items) and 8-40 (1 subscale contains 2 items); higher values represent more quality of life and satisfaction, subscales are summed to combine for total score.
Change in Scales of Psychological Well-being-short form (from baseline to 10-15 weeks post baseline, 6-month follow-up and 12-month follow-up) | Baseline, 10-15 weeks post baseline, 6 and 12 months follow-up
  Self report. Scales of Psychological Well-being-short form: to assess psychological wellbeing; total scores from 1-108, subscales from 1-54; higher values represent more psychological wellbeing; 2 subscales are analyzed separately and not combined.

CONTACTS AND LOCATIONS:
Overall Officials: Brian D. Ostafin, Principal Investigator — University of Groningen
Locations (1):
- Lentis Psychiatric Institute, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vollbehr NK, Hoenders HJR, Bartels-Velthuis AA, Nauta MH, Castelein S, Schroevers MJ, Stant AD, Albers CJ, de Jong PJ, Ostafin BD. Mindful yoga intervention as add-on to treatment as usual for young women with major depressive disorder: Results from a randomized controlled trial. J Consult Clin Psychol. 2022 Dec;90(12):925-941. doi: 10.1037/ccp0000777. PMID 36701531
- See also: Study website with information — http://www.yogabijdepressie.nl